CLINICAL TRIAL: NCT07092488
Title: Application of Platelet-Rich Fibrin (PRF) in Revascularisation of Immature Permanent Teeth
Brief Title: Application of Advanced Platelet-Rich Fibrin Plus (A-PRF+) in Revascularisation of Necrotic Immature Permanent Teeth
Acronym: A-PRF+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Dubravka Turjanski, Dr. Dent. Med., Dr. Dent. Med., University of Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRF-CT-01
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Necrotic Immature Permanent Teeth; Regenerative Endodontic Treatment; Pulp Regeneration; Root Maturation; Periapical Lesions
Keywords: Advanced platelet-rich fibrin; Regenerative endodontics; Immature permanent teeth; Apexification; Calcium hydroxide; Dental pulp regeneration; Revascularization; Platelet-rich fibrin; Advanced platelet-rich fibrin plus
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-group interventional study evaluating the regenerative effectiveness of an advanced platelet-rich fibrin plus (A-PRF+) revascularization protocol in necrotic immature permanent single-rooted teeth. Participants receive the A-PRF+ treatment without randomization or concurrent control groups. The control comparison is conducted retrospectively using historical patient records treated with calcium hydroxide apexification.
Masking Description: While this is an open-label trial with no masking of participants, care providers, investigators, or outcome assessors, radiographic images were randomly coded and evaluated by blinded independent examiners to reduce measurement bias and improve objectivity. Additionally, the control group consisted of randomly selected historical patient records to enhance the validity of comparisons. Follow-up assessments were conducted by independent clinicians who were not involved in the initial treatments, further minimizing examiner bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced Platelet-Rich Fibrin Plus (A-PRF+) Revascularization Group (Experimental): Participants receive the advanced platelet-rich fibrin plus (A-PRF+) revascularization protocol. This involves minimal mechanical instrumentation, canal disinfection with sodium hypochlorite, intracanal medicaments including calcium hydroxide and triple antibiotic paste, followed by placement of autologous A-PRF+ scaffold extending into the coronal cavity. The cavity is then permanently sealed with glass ionomer cement.
  Interventions: Procedure: Advanced Platelet-Rich Fibrin Plus (A-PRF+) Revascularization Procedure

INTERVENTIONS:
Procedure: Advanced Platelet-Rich Fibrin Plus (A-PRF+) Revascularization Procedure — The intervention consists of the advanced platelet-rich fibrin plus (A-PRF+) revascularization protocol. It includes minimal mechanical instrumentation of the root canal, disinfection using sodium hypochlorite irrigation, and intracanal medicaments-initially calcium hydroxide followed by triple antibiotic paste. Peripheral venous blood was drawn from each participant into anticoagulant-free sterile tubes. The blood was immediately centrifuged at 1300 rpm for 8 minutes to obtain the A-PRF+ clot, which was then used as the scaffold material, extending through the root canal into the coronal cavity. The cavity was permanently sealed with glass ionomer cement. This protocol aims to promote regenerative healing and continued root development in necrotic immature permanent teeth.
  Other Names: Advanced platelet-rich fibrin; A-PRF+ revascularization; Platelet-rich fibrin scaffold; Regenerative endodontic procedure with PRF

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of an advanced platelet-rich fibrin plus (A-PRF+) revascularization procedure to promote healing and root development in necrotic immature permanent single-rooted teeth in children and adolescents aged 8 to 18 years.

The main questions it aims to answer are:

* Does the A-PRF+ protocol improve root length, dentinal wall thickness, and apical closure compared to traditional calcium hydroxide apexification treatment?
* Does A-PRF+ promote restoration of pulp vitality and reduce clinical symptoms such as pain, inflammation, or tooth discoloration? Results from the A-PRF+ treatment group will be compared with those from a historical control group receiving traditional calcium hydroxide apexification to evaluate relative effectiveness.

Participants will:

* Receive treatment following the A-PRF+ protocol, which includes disinfecting the tooth canal, applying an autologous platelet-rich fibrin scaffold, and sealing with glass ionomer cement;
* Undergo clinical and radiographic follow-up visits at 1, 3, 6, 9, and 12 months;
* Have pulp vitality tested with cold, electric, and laser Doppler flowmetry methods;
* Be monitored for clinical symptoms, healing progress, and restoration performance.

This study will help determine whether A-PRF+ is a safe and effective alternative to conventional apexification for regenerating necrotic immature teeth in young patients.

DETAILED DESCRIPTION:
This study is a prospective interventional clinical trial evaluating an advanced platelet-rich fibrin plus (A-PRF+) revascularization protocol compared to a historical control group treated with traditional calcium hydroxide apexification for necrotic immature permanent single-rooted teeth in children and adolescents aged 8 to 18 years.

The main goal is to assess the regenerative effectiveness of the A-PRF+ protocol in promoting root development, including root lengthening, dentinal wall thickening, and apical closure, compared to conventional apexification. Secondary objectives include evaluating pulp vitality restoration and monitoring clinical outcomes such as symptom resolution, tooth survival, and adverse effects like tooth discoloration.

Participants in the experimental group were prospectively enrolled and received treatment involving minimal mechanical instrumentation, canal disinfection with sodium hypochlorite, intracanal calcium hydroxide medicament, followed by triple antibiotic paste. At the final appointment, autologous A-PRF+ was prepared from peripheral blood and applied as an intracanal scaffold extending into the coronal cavity, sealed permanently with glass ionomer cement.

The control group consists of patients previously treated at the same institution with calcium hydroxide apexification. Their clinical and radiographic records were retrospectively reviewed for comparison. Apexification was not performed as part of this study.

Clinical and radiographic follow-ups were conducted at 1, 3, 6, 9, and 12 months, including pulp vitality testing with cold, electric, and laser Doppler flowmetry methods, along with standardized periapical radiographs to measure root length, dentinal wall thickness, and apical diameter. Restoration quality was assessed using modified USPHS criteria.

This study aims to determine if the A-PRF+ protocol provides a safe and effective regenerative alternative to traditional apexification for treating necrotic immature teeth, potentially enhancing long-term tooth preservation in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8 to 18 years presenting with immature permanent single-rooted teeth with necrotic pulp caused by caries or dental trauma
* Preserved tooth crown
* Negative response to cold and electric pulp tests
* Radiographic evidence of incomplete root development (Cvek stages I-IV)
* Apical diameter greater than 0.5 mm

Exclusion Criteria:

* Presence of systemic illness or allergies to treatment components
* Complicated crown or root fractures
* Evidence of ankylosis or root resorption
* Ongoing orthodontic treatment
* Inability to comply with follow-up appointments (e.g., needle phobia or poor cooperation)
* Subsequent trauma to the treated tooth during the study period
* Missed recall appointments

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Root Lengthening | From enrollment through 12 months post-treatment
  Root lengthening was assessed by measuring the linear distance from the cementoenamel junction (CEJ) to the radiographic apex on standardized periapical radiographs. Radiographs were obtained using a film holder to ensure consistent angulation and minimize distortion. Measurements were performed using diagnostic software with a precision of 0.1 mm by two independent blinded examiners. The change from baseline to follow-up measurements over the 12-month period was calculated to quantify root lengthening.
Dentinal Wall Thickening | From enrollment through 12 months post-treatment
  Dentinal wall thickening was evaluated by measuring the increase in dentinal wall width at the coronal two-thirds of the root on standardized periapical radiographs. Radiographs were obtained using a film holder to ensure reproducible angulation and reduce distortion. Two blinded examiners independently performed measurements using diagnostic software with an accuracy of 0.1 mm. The difference between baseline and follow-up measurements over 12 months quantified dentinal wall thickening.
Apical Closure | From enrollment through 12 months post-treatment
  Apical closure was assessed by measuring the reduction in apical diameter on standardized periapical radiographs. Radiographs were consistently acquired using a film holder to minimize angulation differences and distortion. Two independent blinded examiners used diagnostic software with 0.1 mm precision to measure the distance across the apical foramen. Changes from baseline to follow-up at 12 months were used to quantify apical closure.

SECONDARY OUTCOMES:
Pulp Vitality Responses | From enrollment through 12 months post-treatment
  Pulp vitality was assessed at each follow-up visit using cold testing and electric pulp testing on the treated tooth and contralateral control tooth. Laser Doppler flowmetry was performed once per patient at either the 9- or 12-month recall to quantitatively measure pulpal blood flow, indicating revascularization. All tests were performed by clinicians blinded to treatment allocation, with responses recorded as positive or negative.
Presence of Periapical Pathology | From enrollment through 12 months post-treatment
  Presence or absence of periapical lesions was evaluated on standardized periapical radiographs at baseline and follow-up visits. Two blinded examiners independently assessed images for periapical pathology. Changes in lesion presence were recorded throughout the 12-month follow-up.
Tooth Survival | From enrollment through 12 months post-treatment
  Tooth survival was defined as retention of the treated tooth throughout the 12-month follow-up period. Any tooth loss or extraction was recorded as an event. Survival status was assessed during clinical recall visits.
Clinical Evaluation of Restorations Using Modified USPHS Criteria | From enrollment through 12 months post-treatment
  Clinical performance of glass ionomer cement restorations was assessed at each recall visit using Modified United States Public Health Service (USPHS) criteria. Parameters evaluated included retention, marginal discoloration, anatomic form, marginal adaptation, secondary caries, and surface texture. Each parameter was scored as Alpha (clinically excellent), Bravo (clinically acceptable), or Charlie (clinically unacceptable/failure).

OTHER OUTCOMES:
Adverse Clinical Events | From enrollment through 12 months post-treatment
  Adverse clinical events including tooth discoloration, abnormal mobility, inflammation, swelling, or sinus tract formation were recorded during clinical examinations at each follow-up visit. All findings were documented in patient records.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric and Preventive Dentistry, University Hospital Centre Zagreb, Zagreb, Croatia, Croatia